CLINICAL TRIAL: NCT05600374
Title: Brain-Oscillation-Synchronized Stimulation to Enhance Motor Recovery in Early Subacute Stroke
Acronym: Boss-Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BOSS-STROKE; CIV-22-01-038788 (Other: EUDAMED-No); 01KG2125 (Other: German Federal Ministry of Education and Research, BMBF)
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled double-blind three-arm parallel-group exploratory clinical trial Medical Device Regulation (MDR) clinical trail
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is a multicenter randomized controlled double-blind three-arm parallel-group exploratory clinical trial. The subjects as well as the as the rater in the post- and the follow-up assessment will be blinded to the intervention condition the patient receives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized stimulation (Experimental): Each 100 Hz triplet is triggered when a real-time analyzed EEG-defined state of high corticospinal excitability is detected (i.e., the negative peak of the ongoing sensorimotor ~10 Hz μ-oscillation).
  Interventions: Device: Bossdevice
- Non-personalized stimulation (No Intervention): The identical rTMS protocol as in Arm 1, but 100 Hz triplets are not synchronized to the ongoing sensorimotor μ-oscillation.
- Sham stimulation (No Intervention): The same protocol as in arm 1 synchronized to the EEG-defined high excitability state, but with ineffective rTMS, using the sham side of an active/placebo TMS coil designed for double-blind clinical trials. Conditions/arm 2 and 3 are control conditions. Arm 2 controls for the specific effect of Condition/arm 1 to synchronize stimulation to the ongoing μ-oscillation. Arm 3 tests if auditory or somatosensory inputs (which are identical in the real and sham stimulation conditions) synchronized with the ongoing μ-oscillation are relevant for the effects of Arm 1.

INTERVENTIONS:
Device: Bossdevice — The bossdevice is a real-time digital signal processor consisting of hardware and software algorithms. It is designed to read-in a real-time raw data stream from a bio-signal amplifier (electroencephalography, EEG), to continuously analyze this data and to detect patterns based on oscillations in different frequencies. When such a specific bio-signal pattern is detected, the device indicates this through a standard output port. This enables a connected device to know with millisecond accuracy when a specific biosignal pattern occurs.
  Arms: Personalized stimulation

SUMMARY:
We will investigate the therapeutic efficacy of EEG-synchronized noninvasive repetitive transcranial magnetic stimulation (rTMS) in the early subacute phase after ischemic stroke to improve upper limb motor rehabilitation. We hypothesize that synchronization of rTMS with the phase of the ongoing sensorimotor oscillation indicating high corticospinal excitability leads to significantly stronger improvement of paretic upper limb motor function than the same rTMS protocol non-synchronized to the ongoing sensorimotor oscillation or sham stimulation.

DETAILED DESCRIPTION:
High-frequency rTMS will be applied to the ipsilesional motor cortex in 400 bursts of 100 Hz triplets with a mean inter-burst interval of 3 s (20 min treatment duration, 1,200 pulses per day) for 5 consecutive workdays (6,000 pulses total) at a stimulus intensity of 80% of resting motor threshold, in one of three conditions/arms, followed by 40 min task-specific hand/arm-physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for admission to the trial:

1. Age ≥ 18 years at the time of signing the informed consent.
2. Cerebral ischemia identified by brain imaging (cerebral MRI or CT) occurred 1-14 days ago.
3. Subject understands and voluntarily signs an informed consent document prior to any study related assessments/procedures.
4. Stroke has resulted in a new arm-/hand motor deficit with ≤ 50 points in the FMA-UE.
5. Presence of motor evoked potentials (MEPs) in the paretic hand. MEPs has to be obtained in the resting muscle

   o If no MEPs can be obtained, MEP search procedure can be repeated later up to 14 days after stroke onset.
6. ● μ-oscillation (8-12 Hz) is recordable by EEG in the ipsilesional sensorimotor cortex with a sufficient signal-to-noise ratio of at least 3 dB
7. ● Subject is able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

Subjects presenting with any of the following criteria will not be included in the trial:

1. Hemorrhagic stroke (this refers to primary intracerebral hemorrhage only; hemorrhagic transformation of ischemic infarcts is not an exclusion criterion)
2. Estimated life expectancy < 12 months
3. Presence of intracranial ferromagnetic metal (extracranial stents ≥10 cm away from the TMS coil are acceptable) in accordance with current safety guidelines [18]
4. Intraocular metal, cochlear implants
5. If TMS might interact with sensors of active implants (e.g., intra-cardiac defibrillators).
6. If a cranial bone gap affects currents induced by TMS (such as after craniotomy).
7. History of seizures or epilepsy.
8. Treatment intervention can't be started within 14 days after onset of stroke.
9. Women during pregnancy and lactation.
10. Participation in other studies if they are MDR or AMG studies or there is otherwise a high risk of insurance law issues intervening between two studies. In case of uncertainty, competing insurances must be contacted prior to participation
11. persistent addiction disorder (except for nicotine dependence)
12. CNS malignoma
13. If there is any concern by the investigator regarding the safe participation of the subject in the study or for any other reason the investigator considers the subject inappropriate for participation in the study.
14. The ability to consent for patients who are unable to speak will be assessed on the basis of the NIHS-Score by an independent physician (details see chapter 21 and appendix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Motor performance after the intervention | After the last treatment session (5 days after first treatment)
  Primary efficacy endpoint is the motor performance after the intervention, as assessed by the Fugl-Meyer assessment (FMA-UE, range 0-66, 0 = no motor function, 66 = normal motor function) of the upper extremity (FMA-UE). The upper-extremity (UE) portion of the Fugl-Meyer assessment is the most frequently used scale to quantify post-stroke motor recovery of the upper extremity. The FMA-UE was used as an endpoint in most of the recent high-frequency rTMS trials in early subacute stroke patients.

SECONDARY OUTCOMES:
Motor performance after 3 months | 3 months after the intervention
  Motor performance 3 months after the intervention, as assessed by the FMA-UE
grip strength | At screening and after 3 months after treatment
  Relative grip strength measured with a vigorimeter (measured in kg).
Assessment to measure quality of life | At screening and after 3 months after treatment
  Stroke-Specific Quality-of-Life Scale (SS-QOL)
modified Rankin Scale Score | At screening and after 3 months after treatment
  Rankin Scale Score (range 0-6, 0 = no disability, 6 =death)
Barthel Index | At screening and after 3 months after treatment
  Barthel Index (ordinary scale ordinal scale 0-100, 0 = fully dependent, 100 =independent in feeding, walking and grooming)
inpatient/npatient rehabilitation | At screening and after 3 months after treatment
  * Number of days as an inpatient (in days)
  * Number of days in inpatient rehabilitation (in days)

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (7):
  - Uniklinik Köln, Klinik und Poliklinik für Neurologie, Cologne
  - Universitätsklinikum Frankfurt, Zentrum der Neurologie und Neurochirurgie, Frankfurt a.M.
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Neurologie, Greifswald
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Neurologie, Leipzig
  - Universitätsmedizin Mainz, Klinik und Poliklinik für Neurologie, Mainz
  - Universitätsklinikum Münster, Klinik für Allgemeine Neurologie, Münster
  - Universitätsklinikum Tübingen, Klinik für Neurologie, Tübingen

REFERENCES:
- [Derived] Lieb A, Zrenner B, Zrenner C, Kozak G, Martus P, Grefkes C, Ziemann U. Brain-oscillation-synchronized stimulation to enhance motor recovery in early subacute stroke: a randomized controlled double-blind three- arm parallel-group exploratory trial comparing personalized, non- personalized and sham repetitive transcranial magnetic stimulation (Acronym: BOSS-STROKE). BMC Neurol. 2023 May 25;23(1):204. doi: 10.1186/s12883-023-03235-1. PMID 37231390